CLINICAL TRIAL: NCT01678703
Title: Randomized Controlled Study: Comparison of Laminaria and Misoprostol for Cervical Preparation Before Second Trimester Surgical Abortion
Brief Title: Comparison of Laminaria and Misoprostol for Cervical Preparation Before Second Trimester Surgical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2trimabort.CTIL
Record Dates: First submitted 2012-08-22; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-07

CONDITIONS: Induced; Abortion, Nonmedical
Keywords: late abortion; laminaria; Misoprostol; Cervical preparation
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laminaria group (Active Comparator): Patients in this group will have cervical preparation with laminaria MedGyn Products, Inc. USA overnight the day before the abortion
  Interventions: Device: Laminaria, MedGyn Products, Inc. USA.
- Misoprostol group (Active Comparator): Patients in this group will have cervical preparation with vaginal Misoprostol 600 mcg overnight the day before the abortion
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Device: Laminaria, MedGyn Products, Inc. USA. — Insertion of Hygroscopic laminarias into the cervical canal for preparation prior to late surgical abortion. The number of laminarias is according to the cervical compliance.
  Other Names: laminaria tents
  Arms: Laminaria group
Drug: Misoprostol — Cervical preparation with vaginal Misoprostol 600 mcg overnight the day before the abortion
  Other Names: Cytotec
  Arms: Misoprostol group

SUMMARY:
This study compares the effectiveness of cervical preparation before second trimester abortion using laminaria versus vaginal Misoprostol.

The investigators hypothesize that medical preparation of the cervix with vaginal Misoprostol is superior to mechanical preparation using laminaria.

The investigators believe that medical preparation makes the procedure easier to perform, equally safe, without addition of pain or discomfort.

DETAILED DESCRIPTION:
This is a prospective randomized study.

The aim of the study is to compare preparation of the cervix before surgical abortion with laminaria and misoprostol.

Primary outcome measures will include:

Initial cervical opening and the need for further dilatation at the procedure Procedure duration

Difficulty score performing the abortion

Complications during and after the procedure

Assessment of pain, using VAS scale, and the need for analgesia before and after the procedure

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients with a viable singleton
* Pregnancy 14-20 weeks of gestation
* Admitted for termination of pregnancy

Exclusion Criteria:

* Contraindication for administration of Misoprostol
* Patients with more than one previous cesarean section scar
* Patients with impaired coagulation
* Significant pulmonary or cardiac disease
* Non viable pregnancy
* Placenta accreta or previa by ultrasound

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2007-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Initial cervical opening and the need for further dilatation at the start of the procedure | 8-12 hours after insersion of laminaria or Misoprostol
  The surgical abortion will be performed 8-12 hours after the insertion of laminaria, or after vaginal application of Misoprostol

SECONDARY OUTCOMES:
pain score during cervical preparation and after the procedure | at the time of the insertion, immediately before the abortion and immediately upon recovery from anesthesia
  The pain score will be accessed immediately after the insertion of the laminaria or the vaginal Misoprostol.
  Pain score will be recorded again right before performing the abortion and will address the 8-12 hours elapsed from the insertion.
  Another assessment of pain will be recorded immediately after the abortion following recovery from general anesthesia

OTHER OUTCOMES:
The degree of difficulty to accomplish the abortion | at the time of performing the surgical abortion
  The difficulty score will be recorded by the surgeon at the operating room immediately upon completion of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Sagiv, MD, Study Director — Tel Aviv University, Sackler Medical School, Israel
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel